CLINICAL TRIAL: NCT06672380
Title: The Influence of Physical Activity on Physical and Emotional Health Indicators in Women Who Have Survived Breast Cancer
Brief Title: The INFLUENCE of PHYSICAL ACTIVITY on the HEALTH and WELL-BEING of BREAST CANCER SURVIVORS
Acronym: PAF-SBM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Bahia (Other)
Responsible Party: Principal Investigator, DARIO DA SILVA MONTE NERO, Master of Science, Federal University of Bahia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 001-PAF-SBM-2024
Record Dates: First submitted 2024-10-31; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer Survivor
Keywords: Breast cancer; Physical exercise; Physical activity; Quality of life; Perceived stress; Sleep quality
MeSH Terms: conditions — Breast Neoplasms; Motor Activity; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Structured and remotely guided physical exercise program for women who are breast cancer survivors (Experimental): Structured and remotely guided physical exercise program The participants in this group took part in a remote exercise program for 3 months, with three classes a week, each lasting 1 hour on alternate days. This group had a more active follow-up, with personalized instruction and ongoing support to improve their physical and emotional health.
  Interventions: Other: Remote Physical Exercise Program for Breast Cancer Survivors
- Initial Consultation and Exercise Guidance via Ebook for Women Surviving Breast Cance (Active Comparator): Arm 2: Initial Consultation and Exercise Guidance via Ebook The participants in this group received an initial consultation, where they were presented with health guidelines and an eBook containing information and guidance on physical exercise. After 30 days, they were given additional encouragement via text message to reinforce physical activity through the eBook, but there was no ongoing direct interaction.
  Interventions: Other: Initial Consultation and Exercise Guidance via Ebook for Women Surviving Breast Cance
- Initial Incentive for Eating Habits in Women Surviving Breast Cancer (Placebo Comparator): Arm 3: The control group only received general guidance on the importance of regular physical activity. The recommendations followed health guidelines, suggesting between 150 and 300 minutes of moderate-intensity physical activity per week.
  Interventions: Other: Initial Incentive for Eating Habits in Women Surviving Breast Cancer

INTERVENTIONS:
Other: Remote Physical Exercise Program for Breast Cancer Survivors — Structured and remotely guided physical exercise program The participants in the intervention group took part in a remote physical exercise program for 12 weeks. The telepresence sessions, conducted three times a week via Google Meet®, lasted 60 minutes and consisted of three phases: warm-up (10 minutes), multi-joint functional exercises (40 minutes) and stretching (10 minutes). The exercises were progressively intensified over the weeks, using the Borg scale to monitor effort. The intensity was adjusted in three cycles: in the first 4 weeks (60 seconds of exercise/90 seconds of rest), in weeks 5 to 8 (75 seconds of exercise/60 seconds of rest) and in weeks 9 to 12 (90 seconds of exercise/30 seconds of rest).
  Other Names: Online Fitness Training for Female Cancer Survivors; Distance Physical Activity Program for Breast Cancer Survivors; Virtual Exercise Intervention for Women Recovering from Cancer; Remote Exercise Classes for Breast Cancer Survivors; Remote Fitness Program for Women with Breast Cancer; Structured and remotely guided physical exercise program
  Arms: Structured and remotely guided physical exercise program for women who are breast cancer survivors
Other: Initial Consultation and Exercise Guidance via Ebook for Women Surviving Breast Cance — Participants in the Ebook group received an illustrated manual containing detailed guidelines for practicing simple physical exercises at home, using only their body weight. The manual suggested a frequency of 3 to 5 times a week, with 30 to 60 minutes of activities such as stretching, squats and exercises for the upper and lower limbs. The participants were encouraged to follow these guidelines and, 30 days after receiving the ebook, an additional stimulus was sent by text message, reinforcing the importance of following the protocol.
  Other Names: Initial Consultation and Exercise Guidance via Ebook
  Arms: Initial Consultation and Exercise Guidance via Ebook for Women Surviving Breast Cance
Other: Initial Incentive for Eating Habits in Women Surviving Breast Cancer — The control group only received general guidance on the importance of regular physical activity. The recommendations followed health guidelines, suggesting between 150 and 300 minutes of moderate-intensity physical activity per week.
  Arms: Initial Incentive for Eating Habits in Women Surviving Breast Cancer

SUMMARY:
Introduction: Cancer remains a leading cause of death globally, with breast cancer being the most common type among women worldwide. The risk of breast cancer is influenced by genetic and lifestyle factors. Healthy dietary habits, regular physical activity, and maintaining a healthy body weight not only reduce the risk of primary neoplastic lesions but also help prevent recurrence. Objective: To assess the impact of educational strategies on behavioral changes, health, and quality of life in women following breast cancer treatment. Methods: This randomized intervention study included 32 participants divided into three groups: remote exercise intervention, e-book guidance, and control. The 12-week intervention involved three weekly sessions with a physical educator and a nutritional consultation. Primary outcomes focused on quality of life, sleep quality, and perceived stress, while secondary outcomes assessed clinical data on biochemical markers, blood pressure, morphofunctional parameters (strength, flexibility, cardiorespiratory capacity), and comorbidities. Women who completed initial breast cancer treatment (surgery, chemotherapy, radiotherapy) and voluntarily participated in the lifestyle program were included in the study. Participants were recruited through invitation letters sent to eligible women from an oncology reference clinic in Salvador. At baseline, standardized questionnaires collected sociodemographic data (age, origin, race, education level), clinical information, and lifestyle habits (smoking, alcohol consumption). Specific questionnaires gathered details on physical activity level (IPAQ), quality of life (SF-36), perceived stress (PSS), sleep quality (PSQI), and morphofunctional assessments (strength tests, BMI, and waist circumference). The questionnaires were administered in person, along with assessments of anthropometric data (BMI, waist circumference), upper and lower limb strength (dynamometry and chair-stand test), cardiorespiratory fitness test, standardized questionnaires, and a 24-hour dietary recall (R24h). Additionally, protocols such as IPAQ, SF-36, PSS, PSQI, and dietary quality questionnaires were used. Intervention: The study intervention focused on developing knowledge about healthy lifestyle habits, emphasizing the benefits of dietary and exercise changes, and promoting motivation and self-confidence to sustain health-oriented behavioral changes. This intervention is anticipated to promote improvements in participant health and lifestyle, impacting their physical health and quality of life.

DETAILED DESCRIPTION:
Ethical Considerations To meet ethical standards, this study, commenced after approval by the Ethics and Research Committee of the School of Nutrition at the Federal University of Bahia (ENUFBA) and the participating institution. Eligible patients were invited to sign the Free and Informed Consent Form (ICF) after receiving all relevant project information, especially regarding procedures and methodology.

It is noteworthy that this project has already been approved-approval numbers 3.935.544 from ENUFBA and 4.185.408 from Santo Antônio Hospital/Sister Dulce Social Works. The study was conducted in accordance with all regulatory guidelines and standards for research involving human subjects as outlined in Resolution 466/2012 of the National Health Council. Participation in the research was voluntary, and all patient information will be kept confidential. Patients who chose not to participate in the study protocol will continue to receive medical and nutritional follow-up at the clinic.

ELIGIBILITY:
Inclusion Criteria:

* Had completed breast cancer treatment (surgery, chemotherapy and/or radiotherapy) at least three months previously.
* Had medical clearance to practice physical activity.
* Were interested in voluntarily participating in the protocol.

Exclusion Criteria:

* They had locomotion or joint limitations that could prevent them from exercising.
* Had psychiatric limitations.
* Were pregnant or breastfeeding.
* Had been doing guided physical activity for at least three months prior to the intervention.
* Did not have access to appropriate technology for remote activities.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-01-29 (Actual); Study Completion 2024-01-29 (Actual)

PRIMARY OUTCOMES:
Quality of life | 12 weeks
  Used a questionnaire (Short Form Health Survey, SF-36), internationally recognized, self-administered questionnaire containing 36 items covering eight physical and mental health domains, and two physical and mental summary scales. The raw scores are recorded, then aggregated and transformed into a scale from 0 to 100, and higher scores indicate better health.
Perceived Stress Scale (PSS-10) | 12 weeks
  Perceived Stress Scale (PSS-10)
  The Perceived Stress Scale (PSS-10) was developed in order to identify life experiences linked to emotion, characterizing the level of stress in the last 30 days, and can be used in any individual over the age of 15.
  Validated in Brazil, this scale consists of 10 multiple-choice items referring to the frequency with which individuals perceive certain situations, with answer options ranging from 1 to 5 (1 = never; 2 = almost never; 3 = sometimes; 4 = almost always and 5 = always). Questions 4, 5, 7 and 8 are scored inverted, as follows: 1=4, 2=3, 3=2, 4=1, 5=0 and the others are added directly in a progressive manner. The total of the scale is the sum of the scores of the 10 questions. The total score can vary from 0 to 40 and the higher the score, the greater the perceived stress. For the purposes of analysis in this study, the stress scale can be analyzed as a qualitative variable, with the total score.
Pittsburgh Sleep Quality Index (PSQI) | 12 weeks
  Sleep quality
  This project will use the Pittsburgh Sleep Quality Index (PSQI), an instrument validated and culturally adapted for the Brazilian population, which subjectively assesses the quality of the sleep pattern, in its general aspects, for the last month in adult individuals.
  The PSQI instrument has 10 questions, of which questions 1 to 4 are open-ended and questions 5 to 10 are semi-open-ended, all of which have space to record comments if necessary. The questions are divided into 7 components: 1) subjective quality, 2) latency, 3) duration, 4) habitual sleep efficiency, 5) sleep disturbances, 6) use of sleep medication, 7) daytime sleepiness and daytime disturbances. Each component is scored from 0 to 3, giving a minimum value of 0 and a maximum of 21 points. The scores are classified as follows: 0-5 as good sleep quality, 6-10 as poor quality and 11-21 as sleep disturbance.
Level of Physical Activity (NAF) | 12 weeks
  Level of Physical Activity (NAF) The level of physical activity was identified using the International Physical Activity Questionnaire (IPAQ), short version, made up of seven open questions. This instrument made it possible to measure the amount of time spent on moderate to vigorous physical activity each week, covering different daily contexts such as domestic activities, leisure, work, commuting and periods of inactivity.
  The IPAQ showed good stability and accuracy, making it suitable for epidemiological studies in various age groups, including young people, adults and the elderly.
  For analysis purposes, individuals who performed less than 150 minutes of physical activity per week were classified as inactive and those who performed more than 150 minutes as active, according to the IPAQ guidelines.

SECONDARY OUTCOMES:
Upper limb strength test Palmar pressure | 12 weeks
  Upper limb strength test Palmar pressure
  To assess muscle strength, the handgrip strength test (HGS) will be applied using a Jamar® hydraulic dynamometer. Patients will sit on a chair with their feet flat on the floor and knees positioned at approximately 90 degrees of flexion. The shoulder of the tested limb is adducted, the elbow is flexed 90 degrees and the hand of the non-tested limb is resting on the thigh of the same side. Participants will be asked to squeeze the handle for 3-5 seconds. Participants will perform three tests with each hand. The value used in this study will be the highest value obtained in any hand. Reference values for the dominant and non-dominant sides will be used to evaluate the measured values.
Lower limb strength test (sit and stand). | 12 weeks
  This test, of low complexity in application and execution, analyzes the movement of sitting and standing, common in everyday life, to assess the strength of the lower limbs.
  A watch with a stopwatch and a chair were used. The test lasted 30 seconds, during which the patient had to perform as many repetitions as possible.
  The patient began by sitting upright (without support), with their feet on the floor and arms crossed over their shoulders. The repetitions were counted out loud, considering only the correct executions, in which the individual stood up completely and returned to the chair, avoiding the back rubbing against the backrest. The patient was instructed to avoid sudden movements to prevent impacts.
  The cut-off point for classifying the patient as independent and able to perform basic movements during training was 9 repetitions in 30 seconds.
The Wells Bench Flexibility Test | 12 weeks
  The Wells Bench Flexibility Test is a validated and widely used method for assessing flexibility. It stands out for its simplicity, easy applicability, low cost and quick execution.
  To carry out the test, a mattress, a Wells bench (a wooden box measuring 30x30 cm and 56 cm long, with a tape measure up to 50 cm) and a protocol sheet were used. The assessor positioned the patient sitting on the mat, with her feet resting on the bench and her legs extended. The patient had to flex her trunk, extending her arms with one hand over the other, trying to reach as far as possible. The movement was repeated three times, considering the greatest distance reached.
  The cut-off point was determined according to each patient's age group, classifying flexibility into five levels: poor, below average, average, above average and excellent.
Cardiorespiratory Capacity Test (6 Minute Walk) | 12 weeks
  Cardiorespiratory Capacity Test (6 Minute Walk) The 6-minute walk test (6MWT) was used to assess cardiorespiratory capacity, providing an analysis of the respiratory, cardiac and metabolic systems based on the distance covered in 6 minutes.
  The application took place on a marked course of 20 to 30 meters, where the participants walked for 6 minutes. Peak oxygen volume (VO2) was calculated using a formula that takes into account distance, age, weight, height and pressure rate (PTP).
  Blood pressure was measured before and after the test with a Missouri® sphygmomanometer and stethoscope, and heart rate was monitored with a Polar® device. VO2 max (ml/kg.min) was classified according to validated parameters for females and age groups.
Anthropometric measurements: Weight | 12 weeks
  Weight: Weight was measured on a calibrated Filizola scale with a capacity of 150 kg and a precision of 100 g. The individual, wearing light clothing and barefoot, was positioned in the center of the scale, with their body erect. The variation allowed between measurements was 0.1 kg, and the weight was recorded and repeated.
Anthropometric measurements: Height | 12 weeks
  Anthropometric measurements
  Height: Height was measured using a stadiometer attached to the scale. The assessor ensured that the individual was not wearing any headgear and was barefoot. The individual stood with their feet together and knees extended, resting the back of their head and shoulders on a vertical surface. The reading was recorded and repeated, allowing for a maximum difference of 0.1 cm.
Anthropometric measurements: Waist circumference (WC) | 12 weeks
  Anthropometric measurements
  Waist circumference (WC): Waist circumference was measured using an inelastic tape, with the individual standing upright, with their waist uncovered and abdomen relaxed. The measurement was taken at the midpoint between the last rib and the iliac crest. The tape was adjusted and the reading taken at the end of breathing, with the procedure repeated and an acceptable variation of 0.5 cm.
ESQUADA (Diet Quality Scale) | 12 weeks
  In the survey, ESQUADA was used as a tool to assess the quality of the participants' diet. This 24-question questionnaire, valid for the Brazilian population, captures eating habits and analyzes aspects such as the frequency of meals, the choice of healthy foods and the consumption of industrialized items.
  The questionnaire covers various aspects of the diet, such as the frequency of main meals, the choice of healthy foods and the consumption of industrialized items. The questions were designed to make it easier for participants to understand and self-assess.
  The answers are scored according to specific criteria, resulting in a classification ranging from "Very Bad" to "Excellent". The categories are
  * Very Bad: Several dietary inadequacies.
  * Bad: Several dietary flaws, but some adequate choices.
  * Good: Balanced diet, but with potential for improvement.
  * Very Good: Meets most nutritional recommendations.
  * Excellent: High quality diet, meeting all guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Dario SM Nero, Master, Principal Investigator — Federal University of Bahia
Locations (1):
- School of Nutrition-Universidade Federal da Bahia, Salvador, Estado de Bahia, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Demographic Data: participants' age, ethnicity, marital status, education and income.
  Clinical Data: Information on treatment (type of surgery, chemotherapy, radiotherapy, hormone therapy) and health conditions (presence of diabetes, hypertension, alcohol and tobacco consumption habits).
  Quality of Life Data: Results of quality of life measurements before and after the interventions, covering aspects such as Physical Limitation, Physical Functioning and Emotional Limitations.
  Physical Activity Data: Level of physical activity and participation in the interventions (remote physical activity or e-book guidance).
  Sleep Quality: Information on sleep patterns and the participants' perception of sleep quality.
  Morphofunctional Aspects: Data on upper and lower limb strength, cardiorespiratory capacity (VO2max) and flexibility.
  Perceived stress: Assessments of the level of stress perceived by the participants.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Individual participant data will be available from [10/11/2024], and will remain accessible until [10/12/2025]. During this period, interested researchers will be able to request access to the data and supporting information, which includes data on sleep quality, morphofunctional aspects, perceived stress and other relevant data collected during the study.
Access Criteria: Academic researchers and health professionals who are involved in studies on breast cancer, physical activity or quality of life.
  Research institutions and universities that have approved research protocols.
  What they can access: Authorized researchers will be able to access:
  Participants' demographic data (age, ethnicity, marital status, education and income).
  Information on health and clinical conditions (diagnosis, treatment, comorbidities).
  Results related to quality of life, sleep quality, perceived stress and morphofunctional aspects (muscle strength, VO2max, flexibility).
  How to access: Those interested should:
  Send a formal request by e-mail to [your e-mail or contact address]. Include a description of the research project and how the data will be used. Provide ethical approval, if necessary. Wait for the request to be analyzed and for a confidentiality agreement to be signed, guaranteeing that the data will be used exclusively for research purposes.
URL: https://drive.google.com/file/d/17k5BTkO5v80vDJNiqvUwNxTpdBQjqviN/view?usp=drive_link